CLINICAL TRIAL: NCT04785118
Title: Hyoscine Butyl-bromide Versus Ondansetron for Nausea and Vomiting During Cesarean Section Under Spinal Anesthesia: A Randomized Clinical Trial
Brief Title: Hyoscine Butyl-bromide Versus Ondansetron for Nausea and Vomiting During Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hyoscine vs Ondansetrone
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Vomiting
MeSH Terms: conditions — Vomiting | interventions — Butylscopolammonium Bromide; Ondansetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- buscopan (Active Comparator): Patients will receive IV hyoscine butyl-bromide 20 mg in 2 ml, just before spinal anaesthesia.
  Interventions: Drug: Hyoscine N Butylbromide
- ondansetron (Active Comparator): Patients will receive IV ondansetron 4 mg in 2 ml, just before spinal anaesthesia.
  Interventions: Drug: Ondansetron
- control (Placebo Comparator): Patients will receive 2 ml of IV normal saline as a placebo just before spinal anaesthesia.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hyoscine N Butylbromide — Patients will receive IV hyoscine butyl-bromide 20 mg in 2 ml, just before spinal anaesthesia.
  Arms: buscopan
Drug: Ondansetron — Patients received IV ondansetron 4 mg in 2 ml, just before spinal anaesthesia.
  Arms: ondansetron
Drug: Saline — Patients received 2 ml of IV normal saline as a placebo just before spinal anaesthesia.
  Arms: control

SUMMARY:
overall incidence of intraoperative nausea and vomiting(IONV) during regional anesthesia for cesarean section is extremely variable, up to 80 percent , depending on the anesthetic technique used (spinal, epidural or combined spinal-epidural) and on the preventive and therapeutic measures taken.1 Spinal anesthesia for CS is safe and effective; it is currently the anesthetic technique of choice for elective Cesarean delivery (CD). However, maternal hypotension associated with spinal anesthesia is one of the primary causes of intraoperative nausea and/or vomiting (IONV); this symptom is thought to be caused by cerebral and gut hypoperfusion that stimulate the vomiting centre in the brainstem and cause serotonin release, respectively.2, 3 While bolus dosing of phenylephrine effectively treats maternal hypotension, it does not prevent intraoperative maternal nausea, which may be associated with established hypotension, and this may adversely affect patient satisfaction.4, 5 However, the unopposed vagal activity that occurs with sympathetic block might be another cause of intraoperative nausea and vomiting during spinal anesthesia.6

Both scopolamine and atropine are tertiary amines, which cross the blood-brain barrier with central side effects, such as confusion, sedation, or paradoxical excitation. However, Hyoscine butyl bromide (HBB) has a quaternary ammonium structure that does not cross through the blood-brain barrier and also with lower placental transfer than atropine, making it more suitable for use in pregnancy 7, 8.

Hyoscine Butyl-bromide, also known as scopolamine butyl-bromide and sold under the brand name Buscopan.9 Despite being a quaternary ammonium compound, HBB is still capable of targeting the chemoreceptor trigger zone due to the lack of a well-developed blood-brain-barrier in the medulla oblongata, which potentiates the antiemetic effects that it produces through local action on the smooth muscle of the gastrointestinal tract.10

So, the aim of the current study is to examine the effect of prophylactic use of HBB and Ondansetron to decrease the incidence of intraoperative bradycardia and thus intraoperative nausea and vomiting in parturients undergoing CD under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18-40 years of age,
* American Society of Anaesthesiologists (ASA) classification class I and II
* patients scheduled for elective or semi-elective surgery (category 3 and 4 Caesarean section) under spinal anaesthesia
* Single baby pregnancy of more than 32 weeks

Exclusion Criteria:

* height < 150 or > 180 cm,
* Body mass index (BMI) >35 kg m-2,
* Contraindication or refusal to undergo regional anaesthesia,
* any cardiovascular disease including arrhythmias, Patients on β-adrenergic blockers or any drugs that may alter the normal response to the study drug,
* history of PONV or motion sickness,
* had taken antiemetic medication in the previous week,
* had a history of hyperemesis gravidarum

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
intraoperative nausea and vomiting | intraoperative
  the incidence of intraoperative all emesis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided